CLINICAL TRIAL: NCT00829621
Title: Incisional Vacuum Assisted Closure (IVAC) Device and Its Effect on Implanted Bone Morphogenic Protein (BMP-2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 1097637
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-10

CONDITIONS: Fractures, Closed
Keywords: BMP-2; Incisional Vacuum Assisted Closure (IVAC)
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 75 mmHg suction (Active Comparator): IVAC suction 75 mmHg
  Interventions: Other: 75 mmHg suction
- 125 mmHg suction (Experimental): IVAC suction 125 mmHg
  Interventions: Other: 125 mmHg

INTERVENTIONS:
Other: 75 mmHg suction — Incisional Vacuum Assisted Closure (IVAC) Device, set to 75 mmHg suction throughout the duration of the IVAC use.
  Arms: 75 mmHg suction
Other: 125 mmHg — Incisional Vacuum Assisted Closure (IVAC) Device, set to 125 mmHg suction throughout the duration of the IVAC use.
  Arms: 125 mmHg suction

SUMMARY:
People who have been scheduled for surgery using Bone Morphogenic Protein (called BMP-2) and an incisional vacuum assisted closure device (called IVAC) will be asked to join this study.

The purpose of this study is to see if using the IVAC device removes BMP-2 from the wound. BMP-2 is a protein used by the body to increase bone healing, decrease the need for additional surgery, and reduce infection rates.

The IVAC is a device that involves a foam dressing secured with an adhesive drape to make an airtight seal over a surgical incision. Tubing runs from the foam dressing to a device that uses gentle suction to drain fluid out (like a vacuum). The IVAC stays on for 48-72 hours depending on amount of drainage. The IVAC by itself helps reduce wound swelling and complications (such as infection).

DETAILED DESCRIPTION:
It is hypothesized that the negative pressure associated with an IVAC is not sufficient to remove BMP-2 from a surgical wound.

BMP-2 is commonly used in open tibia fractures at the time of definitive wound closure, and these wounds are prone to increased swelling and wound complications. The recent observation that IVAC decreases wound edema and increases oxygenation has led to their use in such cases. Used in conjunction, it is entirely possible that the negative pressure exerted by the IVAC can remove BMP-2 from surgical site and therefore decreases the effectiveness of BMP-2. We seek to determine if BMP-2 is present in effluent from the IVAC. If in this study the hypothesis is found to be wrong, and BMP-2 is found within the IVAC effluent, we are prepared to proceed with a follow-up study to quantify the BMP-2 removed by the IVAC.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject has tibia fracture requiring treatment with BMP-2
* Subject to have an Incisional Vacuum Closure (IVAC) Device, placed on the skin directly over the BMP-2 implantation site
* Subject/guardian able to provide informed consent

Exclusion Criteria:

* Subject is less than 18 years old
* Subject has a wound at fracture/surgical site that cannot be closed
* Subject/guardian unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D. Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 75 mmHg: IVAC suction 75 mmHg
  75 mmHg suction: Incisional Vacuum Assisted Closure (IVAC) Device, set to 75 mmHg suction throughout the duration of the IVAC use.
- 125 mmHg: IVAC suction 125 mmHg
  125 mmHg: Incisional Vacuum Assisted Closure (IVAC) Device, set to 125 mmHg suction throughout the duration of the IVAC use.
Period: Overall Study
Arm/Group | 75 mmHg | 125 mmHg
Started | 8 | 12
Completed | 4 | 8
Not Completed | 4 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 75 mmHg | 125 mmHg | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (17.5) | 42.1 (16.6) | 43 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Presence of BMP-2 in Effluent Collected in IVAC Canister
Description: Presence of BMP-2 in effluent collected in IVAC canister
Time Frame: 12-hours, 24-hours, 36-hours, and 48-hours after IVAC application
Measure: Number; unit: participants
Arm/Group | 75 mmHg | 125 mmHg
Number analyzed (Participants) | 8 | 12
participants | 6 | 11
Statistical Analysis 1: Comparison: 75 mmHg vs 125 mmHg; Test type: Superiority or Other; p = 0.36, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | 75 mmHg | 125 mmHg
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/12
Other Adverse Events (participants affected / at risk) | 1/8 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mmHg (N=8) | 125 mmHg (N=12)
died secondary to chronic renal failure (Renal and urinary disorders) | 1 | 0
pulmonary embolis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
wound infection (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mmHg (N=8) | 125 mmHg (N=12)
delayed union (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No